CLINICAL TRIAL: NCT01139684
Title: Development of Field Test for Assessing the Human Anaerobic Capability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Prof. Paltiel Weiner, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: HYMC-0014-10
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Exercise test

ARMS (1):
- Exercise (Experimental)
  Interventions: Behavioral: Repeated sprint test

INTERVENTIONS:
Behavioral: Repeated sprint test

SUMMARY:
A test of the validity of repeated sprint test (RST) 4x 30 meters, against the Wingate Anaerobic Test, which is the gold standard for measuring human anaerobic capacity. The following variables will be used: peak power, mean power and fatigue index. In addition, it will be tested against a 50 meter and a 200 meter shuttle run.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Students

Exclusion Criteria:

* Not healthy

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Human anaerobic capacity | Ten weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Telma Yellin High School, Giv‘atayim, Israel